CLINICAL TRIAL: NCT05614206
Title: Biomarkers Trajectories of Early Intervention in Siblings of Children with Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 897
Record Dates: First submitted 2022-11-03; First posted 2022-11-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder; Early Intervention
Keywords: siblings; autism; biomarkers; early intervention
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Toddlers at elevated likelihood of developing autism with autistic signs, with early intervention (Experimental): Toddlers at elevated likelihood of developing autism with clinical autistic signs who receive an early intervention from 18 to 24 months
  Interventions: Behavioral: Behavioral intervention based on Applied Behavior Analysis principles
- Toddlers at elevated likelihood of developing autism with autistic signs, without early intervention (No Intervention): Toddlers at elevated likelihood of developing autism with clinical autistic signs who do not receive an early intervention
- Toddlers at elevated likelihood of developing autism without autistic signs who received monitoring (No Intervention): Toddlers at elevated likelihood of developing autism without clinical autistic signs who only received assessment and monitoring
- Typically developing toddlers who received monitoring (No Intervention): Typically developing toddlers who only received assessment and monitoring

INTERVENTIONS:
Behavioral: Behavioral intervention based on Applied Behavior Analysis principles — Intervention sessions are conducted by licensed therapists with a training in applied behavior analysis or behavior analysts. One-to-one interventions for 3 h/week are carried out over a period of 5 months.
  The intervention focused on two target symptoms, imitation and joint attention, as two of the pivotal skills in early development. Behavior analytic techniques are used, including discrete trial, shaping for positive reinforcement, systematic prompting and fading procedures, and reinforcement procedures, according to the published manual.
  Imitation sessions start with imitation recognition and imitation of familiar actions (gestural and object imitation) and end with the imitation of novel actions. Joint attention evolvs from initiating requests (starting with gaze shift with the child looking away from an interesting object to the adult and back) to coordination of gaze shift, vocalization and gestures through reaching, and pointing and showing behaviors.
  Arms: Toddlers at elevated likelihood of developing autism with autistic signs, with early intervention

SUMMARY:
This project deals with essential challenges in the context of Autism Spectrum Disorder benefiting from a prospective design in childhood, early intervention and a cutting-edge experimental techniques. The present study tests the potential effect of early intervention on neural and behavioral responses in toddlers at elevated likelihood of developing autism (siblings of children with autism) who show clinical autistic signs. Four comparison groups were included in the study: (1) toddlers at elevated likelihood of developing autism with clinical autistic signs who receive early intervention from 18 to 24 months (2) toddlers at elevated likelihood of developing autism with clinical autistic signs who do not receive early intervention (3) toddlers at elevated likelihood of developing autism without clinical autistic signs who only received assessment and monitoring, and (4) typically developing toddlers who only received assessment and monitoring.

This study focuses on social and nonsocial sensory integration skills (measured by electroencephalographic and eyetracking recordings) to identify reliable biomarkers for early detection and intervention of autism during a critical period of development.

The characterization of biomarkers will guide the detection of the most vulnerable children that will benefit from early intervention, with the long-term aim of reducing the impact of autism on the National Health System.

ELIGIBILITY:
Inclusion Criteria:

* Toddlers aged between 18 and 24 months
* Toddlers at elevated likelihood of developing autism, because siblings of children with a diagnosis of autism (for group 1, 2, and 3)

Exclusion Criteria:

* Gestational age <36 weeks and/or birthweight < 2000 grams
* Griffiths general quotient at 18 months < 70
* presence of major complications in pregnancy and/or delivery likely to affect brain development
* presence of neurological deficits, dysmorphic markers, or other medical conditions.

Ages: 18 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2024-09-26 (Actual)

PRIMARY OUTCOMES:
Change of electroencephalographic theta power (theta frequency band) | once at 18 months of age
  Electroencephalographic theta power to synchronous/asynchronous social and nonsocial stimuli will be measured as an index of social and sensory processing in the 4 groups at T0 (18 months) and T1 (24 months). High-density 128 channel is recorded continuously throughout the session
Change of electroencephalographic theta power (theta frequency band) | once at 24 months of age
  Electroencephalographic theta power to synchronous/asynchronous social and nonsocial stimuli will be measured as an index of social and sensory processing in the 4 groups at T0 (18 months) and T1 (24 months). High-density 128 channel is recorded continuously throughout the session
Change of looking behavior (time of fixations to Area of Interests) and pupillometry parameters (pupil diameter) | once at 18 months of age
  Time of fixations (milliseconds) in different Areas of Interests (i.e., month and eyes) and pupil diameters (millimeters) will be recorded and analysed in the 4 groups at T0 (18 months) and T1 (24 months)
Change of looking behavior (time of fixations to Area of Interests) and pupillometry parameters (pupil diameter) | once at 24 months of age
  Time of fixations (milliseconds) in different Areas of Interests (i.e., month and eyes) and pupil diameters (millimeters) will be recorded and analysed in the 4 groups at T0 (18 months) and T1 (24 months)

SECONDARY OUTCOMES:
Change of standardized scores of clinical measures | Twice: at 18 and at 24 months of age
  Standardized scores (i.e., z-scores, T-scores) of clinical tests (Griffiths Scales, Autism Diagnostic Observation Schedule-Second Edition, McArthur Questionnaire Sensory Profile) will be measured and will be correlated with electroencephalographic (theta power) and eyetracking (looking behavior and pupillometry parameters) data

CONTACTS AND LOCATIONS:
Locations (1):
- Associazione La Nostra Famiglia - IRCCS Eugenio Medea, Bosisio Parini, Lecco, Italy

IPD SHARING:
Plan to Share IPD: No